CLINICAL TRIAL: NCT01524796
Title: NEP-TUNE: Neuropathic Pain - Treatment With Pregabalin Under Real-life Conditions In Denmark
Acronym: NEP-TUNE
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081292; NEP-TUNE (Other: Alias Study Number)
Record Dates: First submitted 2011-12-12; First posted 2012-02-02 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2015-03

CONDITIONS: Peripheral Neuropathic Pain
Keywords: Real-life; non-interventional; observational; peripheral neuropathic pain; Lyrica; pregabalin
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with peripheral neuropathic pain treated with Lyrica
  Interventions: Other: No intervention. Non-interventional study

INTERVENTIONS:
Other: No intervention. Non-interventional study — No intervention. Non-interventional study
  Other Names: pregabalin (Lyrica)

SUMMARY:
Observational study to assess the effectiveness and use of pregabalin (Lyrica) in the treatment of patients with peripheral neuropathic pain in real-life daily clinical practice.

DETAILED DESCRIPTION:
General practitioners and specialists participate in the study. When a subject, independently of the study and before consideration for observation in the study has been prescribed pregabalin for treatment of peripheral NeP, the subject can (before first dose of pregabalin is taken) be included in the observational program.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or over.
* Subjects diagnosed with peripheral neuropathic pain.
* Subjects that independently of the study and before consideration for observation in the study have been prescribed pregabalin for treatment of peripheral neuropathic pain either.

  1. for the first time ('first prescription patients') or
  2. that have not used pregabalin within the previous 6 months but are prescribed pregabalin again ('re-treatment patients')
* Subjects that haven't taken the first dose of the prescribed pregabalin yet.

Exclusion Criteria:

* Subjects not consenting to participate.
* Subjects that at study inclusion (baseline) are on treatment with pregabalin for generalized anxiety or epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: When a subject, independently of the study and before consideration for observation in the study has been prescribed pregabalin for treatment of peripheral NeP, the subject can (before first dose of pregabalin is taken) be included in the observational program.
Sampling Method: Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2012-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081292&StudyName=NEP-TUNE%3A%20Neuropathic%20Pain%20-%20Treatment%20with%20Pregabalin%20Under%20Real-life%20Conditions%20in%20Denmark%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin: Participants who were diagnosed with peripheral neuropathic pain and met the usual prescribing criteria for pregabalin (Lyrica) as per the local product information were observed for a period of 3 months.
Period: Overall Study
Arm/Group | Pregabalin
Started | 128
Completed | 100
Not Completed | 28
Not completed — Adverse Event | 13
Not completed — Lack of Efficacy | 3
Not completed — Lost to Follow-up | 1
Not completed — The price | 1
Not completed — Withdrawal by Subject | 4
Not completed — Move | 1
Not completed — Deterioration of pains | 1
Not completed — Gall stone surgery | 1
Not completed — Nervous about confidentiality | 1
Not completed — Switch to carbamazapine | 1
Not completed — Adverse Event and Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least one dose of the drug under study.
Arm/Group | Pregabalin
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Average Pain Level At Month 3 Telephonic Interview
Description: Pain was assessed on an 11-point numeric rating scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Baseline, Month 3 Telephonic Interview
Population: Analysis population included all participants on pregabalin (Lyrica) at three months follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 86
Units on a scale
  Baseline | 6.7 (1.9)
  Change at Month 3 Telephonic Interview | -2.2 (2.5)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.001, paired Wilcoxon signed-rank test

2. Primary Outcome: Change From Baseline In Worst Pain Level At Month 3 Telephonic Interview
Description: Pain was assessed on an 11-point NRS where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Baseline, Month 3 Telephonic Interview
Population: Analysis population included all participants on pregabalin (Lyrica) at three months follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 86
Units on a scale
  Baseline | 8.4 (1.7)
  Change at Month 3 Telephonic Interview | -2.1 (2.7)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test

3. Primary Outcome: Change From Baseline In Least Pain Level At Month 3 Telephonic Interview
Description: as for outcome 2
Time Frame: Baseline, Month 3 Telephonic Interview
Population: Analysis population included all participants on pregabalin (Lyrica) at three months follow-up.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 86
Units on a scale
  Baseline | 4.1 (2.3)
  Change at Month 3 Telephonic Interview | -1.5 (2.5)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.001, Wilcoxon signed-rank test

4. Secondary Outcome: Sleep Interference Scale Score
Description: Sleep Interference was assessed on an 11-point Sleep Numeric Rating Scale (NRS-11) where a score of 0 indicated "pain did not interfere with sleep" and a score of 10 indicated "pain completely interfered with sleep". Here, "n" signifies "Number of participants" for Baseline and Month 3 telephone interview whereas "n" signifies "number of observations" for Month 1, 2 and 3 because a participant could have had multiple visits during Month 1, 2 and 3 as this was a non-interventional study with no scheduled study visits, except Baseline visit and the Month 3 telephone interview.
Time Frame: Baseline, Month 1, 2, 3, Month 3 telephonic interview
Population: Analysis population included all participants on pregabalin (Lyrica) at three months follow-up. For Baseline and Month 3 telephonic interview, "n" signifies those participants who were evaluable for this outcome. For Month 1 to Month 3, "n" signifies number of observations.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 86
Units on a scale
  Baseline (n = 71) | 5.3 (3.2)
  Month 1 (n= 58) | 4.2 (3.1)
  Month 2 (n= 37) | 4.0 (2.8)
  Month 3 (n= 52) | 4.3 (2.9)
  Month 3 telephonic interview (n= 86) | 2.3 (2.4)

5. Secondary Outcome: Number of Participants With Categorical Scores On Patient Global Impression of Change (PGI-C)
Description: PGIC: participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse). Number of participants in each category are reported.
Time Frame: Month 3 telephonic interview
Population: Analysis population included all participants on pregabalin (Lyrica) at three months follow-up.
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 86
Participants
  Very Much Improved | 18
  Much Improved | 35
  Minimally Improved | 26
  No Change | 4
  Minimally Worse | 3
  Much Worse | 0
  Very Much Worse | 0

6. Secondary Outcome: Health-related Quality of Life Scale Score
Description: Health-related Quality of Life was measured using Euro Quality of Life-5 dimensions (EQ-5D) scale. EQ-5D is a standardized generic instrument to assess health-related quality of life on 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The scale rates current participant's health state on a scale from 0 (worst imaginable health state) to 1 (best imaginable health state); higher scores indicate a better health state. Here, "n" signifies "Number of participants" for Baseline whereas "n" signifies "number of observations" for Month 1, 2 and 3 because a participant could have had multiple visits during Month 1, 2 and 3 as this was a non-interventional study with no scheduled study visits, except Baseline visit and the Month 3 telephone interview.
Time Frame: Baseline, Month 1, 2, 3
Population: Safety analysis set included those participants who received at least 1 dose of the drug under study. Here number of participants analyzed "N" signifies those participants who were evaluable for this measure. For Baseline, "n"=those participants who were evaluable for this outcome. For Month 1 to Month 3, "n"=number of observations.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 104
Units on a scale
  Baseline (n= 104) | 0.47 (0.26)
  Month 1 (n= 81) | 0.58 (0.22)
  Month 2 (n= 52) | 0.58 (0.27)
  Month 3 (n= 64) | 0.63 (0.26)

7. Secondary Outcome: Work Productivity and Activity Impairment (WPAI) Questionnaire
Description: WPAI questionnaire assess work productivity and impairment. It is a patient-rated, six-item questionnaire regarding current employment, hours missed and actually worked, and degree to which a specified health problem affected work productivity and regular activities over the past seven days. Subscale scores include Percent work time missed due to pain (PWP), Percent overall work impairment (PWI), Percent work productivity impairment due to pain (PWPI), Percent overall activity impairment (PAI). Each subscale score is expressed as an impairment percentage (0-100) where higher numbers indicate greater impairment and less productivity. Here, "n" signifies "Number of participants" for Baseline whereas "n" signifies "number of observations" for Month 1, 2 and 3 because a participant could have had multiple visits during Month 1, 2 and 3 as this was a non-interventional study with no scheduled study visits, except Baseline visit and the Month 3 telephone interview.
Time Frame: Baseline, Month 1, 2, 3
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 29
Units on a scale
  PWP Baseline (n= 25) | 28.4 (32.9)
  PWP Month 1 (n= 25) | 28.7 (34.7)
  PWP Month 2 (n=12) | 17.8 (38.6)
  PWP Month 3 (n= 18) | 29.9 (41.6)
  PWI Baseline (n= 23) | 70.0 (22.2)
  PWI Month 1 (n= 24) | 58.2 (28.5)
  PWI Month 2 (n=11) | 48.1 (24.0)
  PWI Month 3 (n= 15) | 56.3 (28.9)
  PWPI Baseline (n= 25) | 63.2 (21.5)
  PWPI Month 1 (n= 25) | 52.0 (25.8)
  PWPI Month 2 (n=12) | 45.8 (18.8)
  PWPI Month 3 (n=19) | 48.9 (23.1)
  PAI Baseline (n= 29) | 68.3 (18.3)
  PAI Month 1 (n= 27) | 63.7 (22.2)
  PAI Month 2 (n=13) | 55.4 (17.1)
  PAI Month 3 (n= 23) | 53.0 (22.2)

8. Secondary Outcome: Pregabalin Dose
Description: Here, "n" signifies "Number of participants" for Baseline and Month 3 telephone interview whereas "n" signifies "number of observations" for Month 1, 2 and 3 because a participant could have had multiple visits during Month 1, 2 and 3 as this was a non-interventional study with no scheduled study visits, except Baseline visit and the Month 3 telephone interview.
Time Frame: After Baseline Visit; Prior to Month 1, 2, 3, Month 3 Telephonic Interview; After Month 1, 2, 3, Month 3 Telephonic Interview
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milligram (mg) per day
Arm/Group | Pregabalin
Number analyzed (Participants) | 86
Milligram (mg) per day
  Dose Prior To Visit: Month 1 (n= 64) | 107.4 (112.7)
  Dose Prior To Visit: Month 2 (n= 48) | 123.4 (102.0)
  Dose Prior To Visit: Month 3 (n= 48) | 164.6 (128.7)
  Dose Prior To Month 3 telephonic interview (n=86) | 240.7 (210.4)
  Dose After Visit: Baseline (n=84) | 81.5 (89.1)
  Dose After Visit: Month 1 (n= 64) | 148.4 (144.5)
  Dose After Visit: Month 2 (n= 48) | 145.3 (115.2)
  Dose After Visit: Month 3 (n= 48) | 169.3 (145.3)

9. Secondary Outcome: Number of Participants Using Other Pharmacological Pain Treatments For Peripheral Neuropathic Pain Before Baseline, Month 1, 2, 3 Visit
Description: Pharmacological treatments included tricyclic antidepressants (TCA), gabapentin, non-steroidal anti-inflammatory drugs (NSAIDs), weak opioids, strong opioids, serotonin-norepinephrine reuptake inhibitors (SNRIs), lidocaine or capsaicin patch (L/C) and other (parcetamol containing drugs, xylocain gel or kinin). Participants may have used more than one pharmacological pain treatments and may be presented in more than 1 category.
Time Frame: Before Baseline, Month 1, 2, 3 Visit
Population: Analysis population included all participants on pregabalin (Lyrica) at three months follow-up. Here "n" signifies pharmacological treatments received at the specified time point.
Measure: Number; unit: Participants
Units Other Than Participants: Treatments
Arm/Group | Pregabalin
Number analyzed (Participants) | 86
Number analyzed (Treatments) | 143
Participants
  Before Baseline Visit: No drug treatment (n= 143) | 5
  Before Baseline Visit: TCA (n= 143) | 14
  Before Baseline Visit: Gabapentin (n= 143) | 33
  Before Baseline Visit: NSAIDs (n= 143) | 25
  Before Baseline Visit: Weak Opioids (n= 143) | 35
  Before Baseline Visit: Strong Opioids (n= 143) | 18
  Before Baseline Visit: SNRIs (n= 143) | 6
  Before Baseline Visit: L/C (n= 143) | 1
  Before Baseline Visit: Other (n= 143) | 6
  Before Month 1 Visit: No drug treatment (n= 71) | 23
  Before Month 1 Visit: TCA (n= 71) | 11
  Before Month 1 Visit: Gabapentin (n= 71) | 2
  Before Month 1 Visit: NSAIDs (n= 71) | 5
  Before Month 1 Visit: Weak Opioids (n= 71) | 17
  Before Month 1 Visit: Strong Opioids (n= 71) | 11
  Before Month 1 Visit: SNRIs (n= 71) | 0
  Before Month 1 Visit: L/C (n= 71) | 1
  Before Month 1 Visit: Other (n= 71) | 1
  Before Month 2 Visit: No drug treatment (n= 60) | 14
  Before Month 2 Visit: TCA (n= 60) | 13
  Before Month 2 Visit: Gabapentin (n= 60) | 2
  Before Month 2 Visit: NSAIDs (n= 60) | 4
  Before Month 2 Visit: Weak Opioids (n= 60) | 14
  Before Month 2 Visit: Strong Opioids (n= 60) | 10
  Before Month 2 Visit: SNRIs (n= 60) | 2
  Before Month 2 Visit: L/C (n= 60) | 0
  Before Month 2 Visit: Other (n= 60) | 1
  Before Month 3 Visit: No drug treatment (n= 58) | 12
  Before Month 3 Visit: TCA (n= 58) | 13
  Before Month 3 Visit: Gabapentin (n= 58) | 0
  Before Month 3 Visit: NSAIDs (n= 58) | 4
  Before Month 3 Visit: Weak Opioids (n= 58) | 16
  Before Month 3 Visit: Strong Opioids (n= 58) | 12
  Before Month 3 Visit: SNRIs (n= 58) | 0
  Before Month 3 Visit: L/C (n= 58) | 0
  Before Month 3 Visit: Other (n= 58) | 1

10. Secondary Outcome: Number of Participants Using Other Pharmacological Pain Treatments For Peripheral Neuropathic Pain After Baseline Visit (Concomitant Medication)
Description: as for outcome 9
Time Frame: After Baseline, Month 1, 2, 3 visit
Population: as for outcome 9
Measure: Number; unit: Participants
Units Other Than Participants: Treatments
Arm/Group | Pregabalin
Number analyzed (Participants) | 86
Number analyzed (Treatments) | 112
Participants
  After Baseline Visit: No drug treatment (n= 112) | 25
  After Baseline Visit: TCA (n= 112) | 12
  After Baseline Visit: Gabapentin (n= 112) | 6
  After Baseline Visit: NSAIDs (n= 112) | 16
  After Baseline Visit: Weak Opioids (n= 112) | 24
  After Baseline Visit: Strong Opioids (n= 112) | 17
  After Baseline Visit: SNRIs (n= 112) | 5
  After Baseline Visit: L/C (n= 112) | 0
  After Baseline Visit: Other (n= 112) | 7
  After Month 1 Visit: No drug treatment (n= 70) | 23
  After Month 1 Visit: TCA (n= 70) | 14
  After Month 1 Visit: Gabapentin (n= 70) | 0
  After Baseline Visit: NSAIDs (n= 70) | 1
  After Month 1 Visit: Weak Opioids (n= 70) | 15
  After Month 1 Visit: Strong Opioids (n= 70) | 15
  After Month 1 Visit: SNRIs (n= 70) | 0
  After Month 1 Visit: L/C (n= 70) | 1
  After Month 1 Visit: Other (n= 70) | 1
  After Month 2 Visit: No drug treatment (n= 60) | 13
  After Month 2 Visit: TCA (n= 60) | 15
  After Month 2 Visit: Gabapentin (n= 60) | 1
  After Month 2 Visit: NSAIDs (n= 60) | 4
  After Month 2 Visit: Weak Opioids (n= 60) | 16
  After Month 2 Visit: Strong Opioids (n= 60) | 9
  After Month 2 Visit: SNRIs (n= 60) | 2
  After Month 2 Visit: L/C (n= 60) | 0
  After Month 2 Visit: Other (n= 60) | 0
  After Month 3 Visit: No drug treatment (n= 58) | 13
  After Month 3 Visit: TCA (n= 58) | 13
  After Month 3 Visit: Gabapentin (n= 58) | 0
  After Baseline Visit: NSAIDs (n= 58) | 3
  After Month 3 Visit: Weak Opioids (n= 58) | 15
  After Month 3 Visit: Strong Opioids (n= 58) | 13
  After Month 3 Visit: SNRIs (n= 58) | 0
  After Month 3 Visit: L/C (n= 58) | 0
  After Month 3 Visit: Other (n= 58) | 1

ADVERSE EVENTS:
Description: Reported in the AE section of the study database. Same participant could have had more than 1 Adverse Event.
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/128
Other Adverse Events (participants affected / at risk) | 21/128
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=128)
Sedation (General disorders) | 4
Dizziness (General disorders) | 5
Oedema (General disorders) | 1
Vertigo (General disorders) | 3
Nausea (General disorders) | 3
Increase in weight (General disorders) | 3
Palpitations (General disorders) | 1
Erectile dysfunction (General disorders) | 1
Reduced energy (General disorders) | 1
Anxiety (General disorders) | 1
Depression (General disorders) | 1
Mood (General disorders) | 1
Head ache (General disorders) | 1
Constipation (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.